CLINICAL TRIAL: NCT03326557
Title: Membrane Sweeping Versus Transcervical Foley Catheter for Induction of Labour in Women With Previous Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Yong Soon Leong, Obstetrician and Gynaecologist, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SibuGHO&G/17-001
Record Dates: First submitted 2017-10-22; First posted 2017-10-31 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Labour, Induced; Vaginal Birth After Caesarean
Keywords: Induction of Labour; Previous Caesarean delivery; Foley; Membrane sweeping; Vaginal delivery
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Intervention Model Description: Pregnant women with one previous Caesarean section who are indicated for induction of labour (IOL) and eligible will be recruited in the study.
  Eligible subjects will be randomly assigned to one of the treatment groups below.
  * Group 1: IOL with membrane sweeping
  * Group 2: IOL with transcervical Foley catheter Blocked randomisation, in a block size of 6 and an allocation ratio of 1:1, will be performed using a computer-generated randomisation sequence by Research Randomizer (available online at https://www.randomizer.org/). The allocation assignment indicating "membrane sweeping" or "transcervical Foley catheter" will be sealed in sequentially numbered, opaque envelopes by principal investigator. Envelopes will be kept in a locked box in Labour Ward. When study consent is signed, the next sequential envelope will be taken out from the box and opened to determine allocation.
Masking Description: This is a non-blinded study in which subjects, medical staffs, and investigators are not blinded to group assignment. This is because both IOL methods are distinctly different procedure. However, both intervention arms are considered receiving equal treatment. In term of safety, both membrane sweeping and transcervical Foley catheter are non-pharmacological in nature and thus the risk of scar rupture does not differ in both methods. In term of efficacy, there is no previous study to compare effectiveness between these two methods. Individual studies revealed that membrane sweeping is likely to reduce the need for formal IOL in post-date pregnancy and transcervical Foley catheter could improve cervical favourability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Membrane sweeping (Active Comparator): Membrane sweeping involves the insertion of a digit past the internal cervical os followed by three circumferential passes of the digit causing separation of the membranes from the lower uterine segment. When the cervix is closed, a massage of the cervical surface for 15 to 30 seconds will be performed instead. Membrane sweeping will be undertaken twice a day at 8 to 10 hours apart.
  Interventions: Procedure: Membrane Sweeping versus Transcervical Foley Catheter for Induction of Labour in Women with Previous Caesarean Delivery
- Transcervical Foley catheter insertion (Active Comparator): Transcervical Foley catheter No. 18 F will be inserted under aseptic technique into the endocervical canal surpassed beyond the internal os. The balloon will be inflated with 60 ml of sterile water and the catheter is plastered to patient's thigh with gentle traction. The catheter will be checked for its position and the traction at 6 hours interval. If it were expelled spontaneously, it would not be re-inserted. Otherwise, the catheter will be removed after 24 hours.
  Interventions: Procedure: Membrane Sweeping versus Transcervical Foley Catheter for Induction of Labour in Women with Previous Caesarean Delivery

INTERVENTIONS:
Procedure: Membrane Sweeping versus Transcervical Foley Catheter for Induction of Labour in Women with Previous Caesarean Delivery — Subjects undergoing induction of labour (IOL) will be randomly assigned to two interventional arms (Group 1: membrane sweeping or Group 2: transcervical Foley catheter insertion). Before IOL, modified Bishop score will be assessed for cervical favourability. After 24 hours of IOL, improvement of modified Bishop score will be reassessed. If the cervix is favourable, amniotomy will be performed followed by augmentation with intravenous oxytocin. If the cervix is still unfavourable and amniotomy is impossible, membrane sweeping will be continued for one more day in Group 1 whereas conservative management will be undertaken for one day in Group 2. Suitability for amniotomy will be reassessed on the next day. After amniotomy, subsequent intrapartum management will be based on the hospital protocol. If amniotomy is still impossible after 2 days of IOL, the ward Obstetrician will discuss with women regarding option of Caesarean section.

SUMMARY:
Nowadays, more and more women embark on pregnancy with previous Caesarean scar. One in five pregnancies requires induction of labour. The use of non-pharmacological methods (methods without using medication) has been gaining popularity for women who are not good candidates, such as women with previous Caesarean scar, for an induction with medications such as prostaglandin. Labour induction with prostaglandin carries higher risk of uterine rupture and thus it is not routinely offered to women with previous Caesarean delivery in Sibu Hospital. Non-pharmacological methods of induction of labour appear to be safe in women with previous Caesarean delivery. However, various methods are available and the efficacy among them remain in doubt.

In Sibu Hospital, membrane sweeping, which is a type of non-pharmacological method, is routinely offered to women with previous Caesarean delivery who require induction of labour. However, membrane sweeping may not exert its labour induction effect immediately and the delivery may be delayed by up to 8 days. This may render a proportion of women to resort to repeated Caesarean section for failed induction.

Transcervical Foley catheter insertion is another non-pharmacological methods for labour induction. Foley catheter, which is made from latex rubber, is inserted into the womb. The balloon will be inflated and this put pressure on the cervix and encourages dilatation. This method may successfully stimulates labour and the catheter falls out once the cervix dilates to 3 centimeters.

The benefits of the Foley catheter:

* A favourable and safe option for mothers who are hoping for a vaginal birth after Caesarean. It is estimated that 4-7 in 10 women with previous Caesarean undergoing labour induction with Foley catheter will have successful vaginal births.
* Cause the cervix to mechanically open without involving medication.
* Reduced risk of uterine rupture compared to induction with prostaglandin.
* Less risk of fetal distress compared to induction with prostaglandin.

The risks of Foley catheter:

* Vaginal bleeding (1.8%)
* Pain requiring removal of catheter (1.7%)
* Baby moving from head down to breech (1.3%)
* Fever (1%) which is lower than induction with prostaglandin.
* The risk of uterine rupture is similar to women undergoing spontaneous vaginal birth after Caesarean.

The aim of this study is to compare the effectiveness of two types of non-pharmacological methods, ie. membrane sweeping and transcervical Foley catheter for induction of labour in women with previous Caesarean delivery.

DETAILED DESCRIPTION:
Induction of labour (IOL) is an obstetric intervention to artificially initiate labour before its spontaneous onset. It is undertaken when maternal or fetal risks of continuing pregnancy outweigh the risks of IOL. The methods of IOL include pharmacological method (prostaglandin), mechanical methods (transcervical Foley catheter and laminaria tents) and surgical method (amniotomy). Pharmacological method and mechanical methods are preferred choice for IOL in women with unfavourable cervix. Whereas surgical method is reserved for women with favourable cervix in which membranes are accessible.

With the global rise in Caesarean section, more and more women embark on pregnancy with previous Caesarean scar. It is estimated that one in every four term pregnancies requires IOL. With IOL in previous Caesarean section, the risk of uterine scar rupture with subsequent catastrophic maternal and neonatal outcomes is the greatest concern. Previous influential study highlighted that IOL with prostaglandin conferred the greatest risk of uterine rupture (2.45%) in women with one previous Caesarean delivery. On the other hand, the risks of uterine rupture were lower and comparable among women whose labour induced without the use prostaglandin (0.77%) and women with spontaneous labour (0.52%). Among the various IOL methods, prostaglandin is more likely associated with shorter interval to achieve vaginal delivery and avoidance of oxytocin augmentation. Nevertheless, mechanical methods have lower risk of uterine hyperstimulation but have more risk of infection. As a result, obstetricians are facing dilemma on deciding the safe and effective method of IOL in women with previous Caesarean delivery.

In Sibu Hospital, membrane sweeping is routinely offered to women with previous Caesarean delivery who require IOL. This technique involves the examining finger passing through the cervix to rotate against the wall of the uterus, to separate the chorionic membrane from the decidua, or to massage around the cervix if the os is closed. However, membrane sweeping may not exert its cervical ripening effect immediately and the delivery may be delayed by up to 8 days. This may render a proportion of women to resort to repeated Caesarean section for failed induction. The vaginal birth rates following membrane sweeping in women with unscarred uterus are ranging between 78%-90%. Among women with previous Caesarean delivery undergoing IOL with membrane sweeping, the reported vaginal birth rates were conflicting. A randomised controlled trial by Hamdan et al. showed vaginal birth rate of 56.1%. Another comparative study by Ramya et al. reported much lower vaginal birth rate of 17.3% which could be explained by high rate of Caesarean Section for maternal request in this study. The average intervals from sweeping to labour onset and to delivery were about 2 days and 4 days, respectively. Membrane sweeping did not increase the risk of maternal or neonatal infection, Caesarean section, postpartum haemorrhage and neonatal poor APGAR score, though discomfort during vaginal examination, minor vaginal bleeding and irregular contraction were frequently reported by women undergoing membrane sweeping. No cases of uterine rupture was reported among women with scarred uterus undergoing membrane sweeping.

Pharmacological IOL method involving prostaglandin is avoided in Sibu Hospital in view of higher risk of scar rupture and presence of limited number of consultants to cope with this debilitating event. Non-pharmacological methods of IOL such as Foley catheter, double-balloon catheter, hygroscopic cervical dilator (laminaria tent) etc are known to have lesser risk of scar rupture. Double-balloon catheters are limited in numbers in this hospital and they are costly. Laminaria tent is not available in this hospital. Foley cathter is a consumable item in this hospital and thus is readily available all the time. Compared to double-balloon catheter, Foley catheter has equivalent cervical ripening efficacy and safety profile. In addition, Foley catheter is also cheaper and has shorter induction to delivery interval. All these advantages make Foley catheter an ideal method of IOL for women with previous Caesarean delivery.

Among women with previous Caesarean delivery underlying IOL with transcervical Foley catheter, the reported vaginal birth rates are ranging between 43.5%-71.4%. The retrospective cohort analysis by Bujold et al. compared the risk of uterine rupture among women with previous Caesarean delivery undergoing spontaneous labour, induction by amniotomy with or without oxytocin, or preinduction cervical ripening with transcervical Foley catheter. The rates of uterine rupture were similar among the groups ((1.1% vs 1.2% vs 1.6%, p = 0.81). However, transcervical Foley catheter appeared to be safer than low dose oxytocin infusion for cervical ripening before amniotomy as the latter tended to be associated with risk of uterine scar dehiscence. Another retrospective cohort study done by Gonsalves et al. showed no case of uterine rupture among 68 women with previous Caesarean section undergoing IOL with transcervical Foley catheter insertion.

The transcervical insertion of balloon catheter as a 'foreign material' may theoretically increase the risk of uterine infection. But, the current data available are conflicting. Meta-analysis by Heinemann et al. demonstrated that the Foley catheter was associated with a significantly higher rate of maternal infections, defined as fever, endometritis or chorioamnionitis, compared to the use of prostaglandins or oxytocin for induction of labour (7.6% vs 5%, pooled OR 1.5, 95%CI 1.07-2.09). On the other hand, Cochrane Review concluded that there is no evidence of an increased risk of infectious morbidity with balloon catheters. In the PROBAAT-trial, comparing the Foley catheter with the use of vaginal prostaglandin E2 gel, the rate of intrapartum infection was significantly lower in women with the Foley catheter (1% vs 3%, p = 0.035). Two other trials evaluating labour induction with balloon catheters after rupture of the membranes did not show an increased risk for maternal infection.

Maslovitz et al. reported the rate of vaginal bleeding of 1.8% following transcervical Foley catheter insertion. However, the bleeding was minor with unaltered haemoglobin levels and coagulation profile. There was also no case of cervical tear which might result in postpartum haemorrhage. Besides, risk of change of fetal vertex presentation to breech was reported to be 1.3%. This was probably related to concomitant presence of unengaged free-floating fetus and contraction following Foley catheter insertion which resulted in flipping movement of the fetus. Risk of poor APGAR and NICU admission was not significantly higher compared to other IOL methods eg. prostaglandin and oxytocin.

Till date, there is paucity of evidence on the superiority of membrane sweeping and transcervical Foley catheter in IOL in previous Caesarean delivery. Both methods have the same mechanism action by increasing local production of endogenous prostaglandin. The aim of this study is to evaluate the effectiveness of membrane sweeping and transcervical Foley catheter insertion for IOL in women with previous Caesarean delivery.

The investigators had searched electronic databases including PubMed, Cochrane Library, Scopus, Ovid, JSTOR and Google Scholar. The investigators found that there was no study comparing these two IOL methods, thus no prior information is available for sample size calculation. Based on Julious SA, the investigators recruited 24 subjects (a sample size of 12 per group) from 15 February 2018 to 8 May 2018 and performed an interim analysis to calculate the actual sample size required for a full randomised controlled trial (RCT). The justifications for this interim sample size were based on rationale about feasibility, precision about the mean and variance, and regulatory considerations. The justifications for this interim sample size are based on rationale about feasibility, precision about the mean and variance, and regulatory considerations.

The final sample size was calculated based on the study primary outcome of achievement of favourable cervix (Bishop score of 8 or more) within 48 hours of IOL. From the interim analysis, the investigators found that the rate of favourable Bishop score achieved within 48 hours of IOL was 58.3% for membrane sweeping arm and 91.7% for transcervical Foley catheter arm. The investigators used the following formula by Fleiss JL. 1981 to calculate the final sample size. With α at 0.05 and power at 0.8, total of 52 subjects (26 subject in each arm) need to be recruited. With the estimated dropout rate of 15%, the final sample size required is 60 subjects, which means a further 36 subjects (18 subjects on each arm) will be recruited to complete the study. In addition, data of the initial 24 subjects (12 per arm) recruited will be included in the final data analysis. This further recruitment will not affect the randomisation of the previous and future subjects because blocked randomisation, in a block size of 6 and an allocation ratio of 1:1 is used. Furthermore, there is no change in the methodology, scale and instrument of the research.

The investigators had applied ethical approval of the recruitment of a further 36 subjects from the Malaysia Research and Ethics Committee, Ministry of Heath Malaysia and the application was approved on 12 June 2018.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with one previous Caesarean section who are admitted to Sibu Hospital for induction of labor (IOL) will be recruited. The inclusion criteria are age at least 18 years old, gestational age ≥ 37 weeks, singleton pregnancy, reassuring fetal status and modified Bishop score ≤ 6.

Exclusion Criteria:

* Ruptured membranes, intrauterine death, polyhydramnios, severe fetal anomalies, and multiple pregnancy.
* Contraindications for IOL eg. placenta previa, suspected macrosomia, suspected cephalopelvic disproportion, non-cephalic presentation, and obstructive pelvic masses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Achievement of favourable cervix (Bishop score of 8 or more) within 48 hours of induction of labour | From the time of commencing induction until the time whereby the cervix becomes favourable (Bishop score of 8 or more), assessed up to 48 hours
  The number of subjects who achieve Bishop score of 8 or more within 48 hours of induction of labour

SECONDARY OUTCOMES:
Induction outcomes: Improvement of modified Bishop score at interval of 24 hours after induction | From the time of commencing induction till 24 hours after induction
  The difference of modified Bishop score between pre-induction and 24 hours post-induction. The score is assessed based on the station of the presentation, os dilation, and effacement (or length), position and consistency of the cervix. Score ranges from 0 to 12. A score of 8 or more generally indicates that the cervix is ripe/favourable.
Induction outcomes: Improvement of modified Bishop score at interval of 48 hours after induction | From the time of commencing induction till 48 hours after induction
  The difference of modified Bishop score between pre-induction and 48 hours post-induction. The score is assessed based on the station of the presentation, os dilation, and effacement (or length), position and consistency of the cervix. Score ranges from 0 to 12. A score of 8 or more generally indicates that the cervix is ripe/favourable.
Delivery outcomes: Mode of delivery | At time of delivery
  Final mode of delivery ie. vaginal delivery and Caesarean section
Delivery outcomes: Duration of oxytocin augmentation | From the time of administrating oxytocin augmentation until the time of delivery, assessed up to 16 hours
  Duration of oxytocin augmentation during intrapartum period
Delivery outcomes: Induction to vaginal delivery interval | From the time of induction of labour until the time of vaginal delivery, assessed up to 72 hours
  Duration between the time of induction of labour and vaginal delivery
Delivery outcomes: Amniotomy to vaginal delivery interval | From the time of amniotomy till the time of vaginal delivery, assessed up to 16 hours
  Duration between the time of amniotomy and vaginal delivery
Maternal outcomes: Uterine hyperstimulation | From the time of induction until the time of delivery, assessed up to 72 hours
  The occurrence of uterine hyperstimulation (> 5 contractions per 10 minutes for at least 20 minutes or a contraction lasting at least 2 minutes with/without abnormal fetal heart rate) during labour process
Maternal outcomes: Uterine rupture | From the time of induction until the time of delivery, assessed up to 72 hours
  The occurrence of uterine rupture during labour process
Maternal outcomes: Post-partum haemorrhage | From the time of delivery until the time of discharge, assessed up to 48 hours
  The occurrence of post-partum haemorrhage (estimated blood loss ≥ 500 ml) after delivery
Maternal outcomes: Maternal pyrexia | From the time of induction until the time of delivery, assessed up to 72 hours
  The occurrence of maternal fever (temperature >38.0 °C once, or 37.5 °C on two occasions 2 hours apart) during labour process
Maternal outcomes: Duration of hospitalisation | From the time of induction until the time of discharge home following delivery, assessed up to 120 hours
  To measure the duration of hospitalisation required
Neonatal outcomes: 5-minutes APGAR score | Upon the baby is delivered, assessed up to 5 minutes of life
  To measure the APGAR score of the newborn at 5 minutes of life, scores range between 0 to 10, score < 7 is considered abnormal
Neonatal outcomes: cord pH | Upon baby is delivered, assessed immediately
  To obtain umbilical cord blood of the newborn for pH measurement upon birth, normal levels are 7.25 and above, pH < 7.25 is abnormal and < 7.0 is considered pathological acidosis due to perinatal asphyxia

CONTACTS AND LOCATIONS:
Overall Officials: Soon Leong Yong, MD, Dr. ObGyn, Principal Investigator — Department of Obstetrics and Gynaecology, Sibu Hospital, Sarawak, Malaysia.
Locations (1):
- Sibu Hospital, Sibu, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT03326557/Prot_SAP_ICF_000.pdf